CLINICAL TRIAL: NCT06875362
Title: Safety and Efficacy of LR08 in Modulating Gut Microbiota and Improving Metabolic Health in Healthy Adults: A Clinical Study
Brief Title: Probiotic LR08 Improves Gut and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20250308
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy Adults
Keywords: Probiotics; Efficacy; Safety; Gut Microbiota; Immune Function
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Intervention with probiotic LR08 (30 billion CFU/day, 3g) was administered daily for 8 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Every day to give 3 g maltodextrin intervention for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The trial period of this study lasts for 2 months(8weeks), during which each participant will have 3 visits (at month 0, month 1, andmonth 2).
  Arms: Probiotic group
Dietary Supplement: Placebo — The trial period of this study lasts for 2 months(8weeks), during which each participant will have 3 visits (at month 0, month 1, andmonth 2).
  Arms: Placebo group

SUMMARY:
Evaluate the efficacy and safety of LR08 as a dietary supplement compared to a placebo in enhancing intestinal health and immune function in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to attend 3 follow-up visits during the intervention period
2. Agree to provide blood, urine, and stool samples twice during the intervention period
3. Good eyesight, able to read and write, and capable of wearing glasses if needed
4. Good hearing and able to fully comprehend all instructions during the intervention

Exclusion Criteria:

1. Presence of digestive diseases, particularly gastrointestinal disorders (e.g., celiac disease, ulcerative colitis, Crohn's disease)
2. History of serious neurological conditions (e.g., epilepsy, stroke, severe head trauma, meningitis within the last 10 years, brain surgery, brain tumor, or prolonged coma-not including general anesthesia)
3. History of or currently receiving treatment for mental health disorders such as alcohol/drug/substance abuse, schizophrenia, psychosis, or bipolar disorder
4. Currently taking medication for depression or low mood
5. Presence of internal organ failure (e.g., heart, liver, or kidney failure)
6. History of radiation therapy or chemotherapy treatments
7. Underwent general anesthesia within the past three years or are scheduled for general anesthesia within the next 3 months during the trial period
8. History of hepatitis (B or C), HIV, or syphilis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Immune Function | Week 0 and Week 8
  Evaluation of immune function markers, specifically immunoglobulin A (IgA) concentration, to assess the effects of LR08 supplementation compared to placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Xu fei, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Han M, Xu F, Dong Y, Zhu J, Fang S, Zhao L. Safety and immune-regulating effects of Limosilactobacillus reuteri LR08: Preclinical and clinical evidence from a randomized controlled trial. Clin Nutr. 2026 Jan 20;58:106582. doi: 10.1016/j.clnu.2026.106582. Online ahead of print. PMID 41650801